CLINICAL TRIAL: NCT04605965
Title: Wearable Health Data to Investigate Long-term Cardiovascular and Behavioral Health Outcomes in COVID-19 Patients After Discharge: The WEAICOR Study
Brief Title: WEAICOR: Wearables to Investigate the Long Term Cardiovascular and Behavioral Impacts of COVID-19
Acronym: WEAICOR
Status: Active, not recruiting | Type: Observational
Sponsor: Tulane University (Other)
Collaborators: Biostrap (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-678
Record Dates: First submitted 2020-08-12; First posted 2020-10-28 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Covid19; Cardiovascular Complication; Behavioral Changes
Keywords: Digital Health
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational COVID-19 study that uses wearable health monitoring technology to follow COVID-19 positive individuals to monitor persistent symptoms and any potential long-term complications or cardiovascular and behavioral impacts from the disease.

DETAILED DESCRIPTION:
Participants will wear a Biostrap wristband device that captures high-fidelity, raw photoplethysmography (PPG) waveforms and collects important indicators of heart and mental health, including heart rate, heart rate variability, pulse points, oxygen saturation and sleep patterns. Biometric data will be collected and participants will be alerted if any measurements are outside their normal range.

Researchers are recruiting 200 participants who were diagnosed with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Positive COVID-19 diagnosis
* Ages 18 to 120
* Access to WiFi

Exclusion Criteria:

* Negative COVID-19 diagnosis
* Age younger than 18 and older than 120
* Lack of access to WiFi

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a positive COVID-19 diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of major cardiovascular events | 12 Months
  Including arrhythmia occurrence or recurrence, congestive heart failure, myocardial infarction, cardiomyopathy and ischemic stroke.
Incidence of atrial arrhythmia | 12 Months
  Including atrial fibrillation, atrial flutter, atrial tachycardia
Mental health effect of COVID-19 measured by incidence of Generalized Anxiety Disorder (GAD) using Generalized Anxiety Disorder 7-item (GAD-7) Scale | 12 Months
  Generalized Anxiety Disorder 7-item (GAD-7) Scale includes 7 questions to be answered by the patient, each answer is scored from 0 to 3, and the scale range is from 0 to 21, with a higher number representing more severe GAD level
Mental health effect of COVID-19 measured by incidence of depression using Beck Depression Fast Screen Scale | 12 Months
  Beck Depression Fast Screen Scale includes 21 questions to be answered by the patient scored from 0 to 3, and the scale range is from 0 to above 40, with a higher number representing more severe depression level
Mental health effect of COVID-19 measured by incidence of Post Traumatic Stress Syndrome (PTSD) using the Post Traumatic Stress Disorder Checklist- Standard Form (PCL-S) scale | 12 Months
  Post Traumatic Stress Disorder Checklist- Standard Form (PCL-S) Scale includes 20 questions to be answered by the patient scored from 1 to 5. Total symptom severity score (ranging 0-80) can be obtained by summing the scores for each of the 20 items. Higher number represents more likely that the patient has PTSD.
Mental health effect of COVID-19 measured by incidence of substance abuse using a baseline use of alcohol survey | 12 Months
  Baseline use of alcohol survey includes ten questions to be answered by the patient scored from 0 to 4 with a higher number representing increased alcohol consumption
Mental health effect of COVID-19 measured by incidence of substance abuse using a baseline use of drugs survey | 12 Months
  Baseline use of drugs survey includes ten questions to be answered by the patient scored from 0 to 4 with a higher number representing increased drug use
Mental health effect of COVID-19 measured by incidence of substance abuse using a baseline use of nicotine products survey | 12 Months
  Baseline use of nicotine products survey includes 4 questions to be answered by the patient to find out which nicotine products the patient is using if any and how many cigarettes they're smoking per day

CONTACTS AND LOCATIONS:
Overall Officials: Nassir Marrouche, MD, Principal Investigator — Tulane University School of Medicine
Locations (2):
- United States (2):
  - Tulane University, TRIAD Center, New Orleans, Louisiana
  - Tulane University, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data may be used for secondary analyses/research on COVID19 complications